CLINICAL TRIAL: NCT04236804
Title: VANISH (Virtual Autonomic Neuromodulation Induced Systemic Healing) for Chronic Low Back Pain (CLBP)
Brief Title: VANISH for Chronic Low Back Pain
Acronym: VANISH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ajay Wasan, MD, Msc (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Ajay Wasan, MD, Msc, Professor of Anesthesiology and Perioperative Medicine and Psychiatry, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY19050295; 1R44DA049630-01 (NIH)
Record Dates: First submitted 2019-12-06; First posted 2020-01-22 (Actual); Results first posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-03

CONDITIONS: Chronic Low-back Pain
Keywords: Virtual Autonomic Neuromodulation Induced Systemic Healing; TMC-CP01

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- TMC-CP01 Intervention (Experimental): Ten patients will be randomly assigned to receive the TMC-CP01 intervention every day for 8 weeks in addition to their current opioid prescription and tapering guidelines.
  Interventions: Device: Flowly (TMC-CP01)
- Standard of Care (No Intervention): Ten patients will be randomly assigned to receive their current opioid prescription and tapering guidelines, as standard of care.

INTERVENTIONS:
Device: Flowly (TMC-CP01) — TMC-CP01 is a device designed specifically for pain management and is tailored for low back pain. The treatment utilizes virtual reality and biofeedback to train patients to auto-regulate themselves and improve their pain over time guidelines.
  Other Names: Virtual Reality
  Arms: TMC-CP01 Intervention

SUMMARY:
The program, called TMC-CP01, will use a combination of virtual reality, biofeedback, and psychological exercises to manage pain associated with Chronic Low Back Pain. Chronic pain affects an estimated 100 million Americans, around one-third of the U.S. population. One of the most prevalent conditions under chronic pain is Chronic Low Back Pain (CLBP). About 27% of chronic pain patients experience CLBP. It is the leading cause of disability in the world and 31 million Americans suffer from CLBP. The most common analgesic tool for pain patients, especially for LBP patients, is opioids. However, opioid users are subject to drug tolerance and physical dependence, which decreases efficacy and increases risk of complication. Long-term users often require doses up to ten times their original dose to achieve equivalent analgesia and, after months of exposure, patients' risk of addiction increases.

This project aims to introduce a digital intervention to standard CLBP management with a virtual reality-enabled pain management system that will improve pain management and decrease daily dosages of opioids.

DETAILED DESCRIPTION:
TMC-CP01 is a treatment based on the VANISH (Virtual Autonomic Neuromodulation Induced Systemic Healing) system and method, which combines existing technologies and therapies into Virtual Reality (VR) to help people learn to auto-regulate the way their body feels. TMC-CP01 is designed specifically for pain management and is tailored for low back pain. The treatment utilizes virtual reality and biofeedback to train patients to auto-regulate themselves and improve their pain over time. By providing patients an accessible and effective alternative pain management tool, patients can avoid opioid use, dependency, and resulting complications due to opioids. Change in daily opioid dose, expressed in morphine equivalents, is the primary outcome. TMC-CP01 uses virtual reality as a platform to enable and optimize biofeedback training and psychological exercises.

Virtual Reality, alone is a proven method for pain management both through distraction and through active pain control mechanisms. Due to its stimulating nature, VR has the power to claim the majority of a user's attention and distract them from other stimuli such as pain. Because it is so visually engaging, VR is a powerful tool for visualization, which can be used to optimize and enhance visualization of biofeedback. VR can also affect users' emotions and perception by providing a sense of presence and psychological engagement. With recent developments in portable head mounted display (HMD) technology, VR has become accessible to people on a much broader and more affordable scale and it represents an ideal platform to develop a non-invasive pain management tool for chronic pain. Biofeedback is at the heart of TMC-CP01 and is the main mechanism by which patients learn to control their physiology. By allowing patients to visualize their physiological processes, patients gain a greater mind-body awareness and can learn to auto-regulate physiological functions that previously seemed out of their control.

ELIGIBILITY:
Inclusion Criteria:

* Females or males 18 years of age and older at screening
* Diagnosis of Chronic Lower Back Pain (CLBP) and a >50mg MME daily opioid dosage
* Able to provide informed consent, adhere to the study visit schedule, and complete all study assessments
* Signed informed consent form

Exclusion Criteria:

* Subjects who, in the opinion of the study site principal investigator, have a psychotic disorder, dementia, or other issue which may make accurate data reporting difficult
* Subjects who do not speak fluent English
* Patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-06-17 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Wasan, MD, MSc, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Pain Medicine At Centre Commons, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TMC-CP01 Intervention | Standard of Care
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TMC-CP01 Intervention | Standard of Care | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.70 (14.30) | 58.8 (10.11) | 57.25 (12.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 8 | 12
  Male | 6 | 2 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 9 | 9 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Opioid Use Via Subject Report
Description: Daily dose of oral opioids recorded as morphine equivalents will be collected
Time Frame: Week 0
Measure: Mean (Standard Deviation); unit: morphine milligram equivalent
Arm/Group | TMC-CP01 Intervention | Standard of Care
Number analyzed (Participants) | 10 | 10
morphine milligram equivalent | 47.5 (36.53) | 21.75 (23.19)

2. Secondary Outcome: Assessment of Opioid Use Via Subject Report
Description: The amount and dosing of opioid medications taken by each subject will be recorded throughout the study. The lower the average daily morphine milligram equivalent [MME], the better the outcomes. Outcomes will be measured over the span of the study and compared between the two groups.
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: MME
Arm/Group | TMC-CP01 Intervention | Standard of Care
Number analyzed (Participants) | 10 | 10
MME | 47.27 (36.77) | 10.75 (7.34)

3. Secondary Outcome: Assessment of Opioid Use Via Subject Report
Description: as for outcome 2
Time Frame: Week 8
Measure: Mean (Standard Deviation); unit: MME
Arm/Group | TMC-CP01 Intervention | Standard of Care
Number analyzed (Participants) | 10 | 10
MME | 47.27 (36.77) | 10.62 (7.36)

4. Secondary Outcome: Flowly (TMC-CP01) Virtual Reality Intervention Feasibility Via Change From Baseline in Heart Rate Variability (HRV) at 8 Weeks
Description: HRV will be modulated by conforming respiration and heart rate to optimal breathing patterns. The games are designed to guide subjects' physiology to a more optimal state for pain reduction using biofeedback. Resonant breathing is breathing that activates the coordinated function of oscillating body systems. This breathing increases your Heart Rate Variability. Greater Heart Rate Variability (a higher HRV score) at rest indicates better outcomes. Outcomes will be measured over the span of the study and compared between the two groups.
Time Frame: 8 Weeks
Population: HRV data were not collected due to a malfunction in the Flowly app, which was in beta testing during the study. The app was intended to collect HRV via a paired biometric sensor, but it failed to reliably communicate with the device. As a result, HRV measurements were not transmitted or stored, and no usable data were available for analysis.
Arm/Group | TMC-CP01 Intervention | Standard of Care
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change From Baseline in Opioid Cravings Using the Craving Index at 8 Weeks
Description: The Craving Index questionnaire on the Flowly app assesses opioid cravings using 6 qualitatively scaled questions, ranging from 'none' (minimum score: 0) to 'the greatest possibility' (maximum score: 5 per question, total score: 30). Lower scores indicate less frequent opioid cravings, suggesting better outcomes. Measurements were assessed weekly, and the analysis focused on comparing scores between baseline and 8 weeks to evaluate changes in cravings between the two groups.
Time Frame: weekly, up to 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TMC-CP01 Intervention | Standard of Care
Number analyzed (Participants) | 10 | 10
score on a scale | 0.60 (7.56) | 0.83 (4.92)

6. Secondary Outcome: Change From Baseline in Physical Function Using PROMIS Physical Function Short Form T-score at 8 Weeks
Description: The investigators used the PROMIS Physical Function Short Form T-score to assess key patient-centered outcomes related to physical function. This assessment includes 4 physical function-related questions, each scored on a 5-point Likert scale (1 = unable to do, 5 = without any difficulty). The raw total score ranges from a minimum of 4 to a maximum of 20.
  Responses were converted to T-scores, where the mean in the general population is 50 with a standard deviation of 10. Higher T-scores indicate better physical function, while lower T-scores suggest worse physical function. Clinically relevant thresholds may indicate that lower scores are associated with greater physical disability.
  Measurements were conducted at baseline and Week 8, with the analysis focused on comparing changes in physical function between the two groups.
Time Frame: Assessed weekly, change from baseline and Week 8 reported
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | TMC-CP01 Intervention | Standard of Care
Number analyzed (Participants) | 10 | 10
T-score | 0.07 (2.89) | -1.41 (4.24)

7. Secondary Outcome: Change From Baseline in Fatigue Using PROMIS Fatigue Short Form T-score at 8 Weeks
Description: The investigators used the PROMIS Fatigue Short Form T-score to assess key patient-centered outcomes related to fatigue. This assessment includes 4 fatigue-related questions, each scored on a 5-point Likert scale (1 = not at all, 5 = very much). The raw total score ranges from a minimum of 4 to a maximum of 20.
  Responses were converted to T-scores, where the mean in the general population is 50 with a standard deviation of 10. Higher T-scores indicate greater fatigue, while lower T-scores suggest less fatigue, which reflects better outcomes. Clinically relevant thresholds suggest that elevated T-scores may indicate increased fatigue severity.
  Measurements were conducted at baseline and Week 8, with the analysis focused on comparing changes in fatigue levels between the two groups.
Time Frame: Baseline and Week 8
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | TMC-CP01 Intervention | Standard of Care
Number analyzed (Participants) | 10 | 10
T-score | 0.17 (5.05) | 0.61 (8.09)

8. Secondary Outcome: Change From Baseline in Pain Interference Using the PROMIS Pain Interference Short Form at 8 Weeks
Description: The investigators used the PROMIS Pain Interference Short Form to assess how pain impacts daily activities. This measure includes 5 pain-related questions, each scored on a 5-point Likert scale (1 = not at all, 5 = very much). The raw total score (range: 5 to 25) was converted to a standardized T-score (mean = 50, SD = 10).
  Higher T-scores indicate greater pain interference, while lower T-scores suggest less interference (better outcomes). A T-score of 60+ may indicate clinically significant pain interference, while 40 or lower suggests minimal interference.
  Measurements were conducted over the study, with scores compared between baseline and 8 weeks to assess changes in pain interference.
Time Frame: Assessed weekly, change from baseline and Week 8 reported
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | TMC-CP01 Intervention | Standard of Care
Number analyzed (Participants) | 10 | 10
T-score | -1.47 (3.69) | -1.75 (3.22)

9. Secondary Outcome: Change From Baseline in Pain Intensity Using the PROMIS Pain Intensity Item at 8 Weeks
Description: The investigators used the PROMIS Pain Intensity Item to assess patients' self-reported pain levels. This measure consists of one question, scored on an 11-point Likert scale (0 = no pain, 10 = worst imaginable pain). The raw score was converted to a standardized T-score (mean = 50, SD = 10).
  Higher T-scores indicate greater pain intensity, while lower T-scores suggest less pain (better outcomes). A T-score of 60+ may indicate clinically significant pain, while 40 or lower suggests mild or minimal pain.
  Measurements were conducted throughout the study, with scores compared between baseline and 8 weeks to assess changes in pain intensity.
Time Frame: Assessed weekly, change from baseline and Week 8 reported
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | TMC-CP01 Intervention | Standard of Care
Number analyzed (Participants) | 10 | 10
T-score | 0.2 (1.32) | 0.14 (1.07)

10. Secondary Outcome: Change From Baseline in Sleep Disturbance Using the PROMIS Sleep Disturbance Short Form at 8 Weeks
Description: The investigators used the PROMIS Sleep Disturbance Short Form to assess patient-reported sleep difficulties. This measure includes 4 items, each rated on a 5-point Likert scale (1 = not at all, 5 = very much). The raw score (range: 4 to 20) was converted to a T-score (mean = 50, SD = 10).
  Higher T-scores indicate greater sleep disturbance (worse outcomes), while lower T-scores suggest better sleep quality. A T-score of 60+ may indicate clinically significant sleep disturbance, while 40 or lower suggests minimal issues.
  Measurements were conducted throughout the study, with scores compared between baseline and 8 weeks to assess changes in sleep disturbance.
Time Frame: Assessed weekly, change from baseline and Week 8 reported
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | TMC-CP01 Intervention | Standard of Care
Number analyzed (Participants) | 10 | 10
T-score | -1.82 (5.73) | -0.47 (4.51)

11. Secondary Outcome: Change From Baseline in Ability to Participate in Social Roles and Activities Using the PROMIS Short Form at 8 Weeks
Description: The investigators used the PROMIS Ability to Participate in Social Roles and Activities Short Form to assess social participation. This measure includes 4 items, each rated on a 5-point Likert scale (1 = never, 5 = always). The raw score (range: 4 to 20) was converted to a T-score (mean = 50, SD = 10).
  Higher T-scores indicate greater ability to engage in social roles and activities (better outcomes), while lower scores suggest more social restrictions. A T-score below 40 may indicate clinically significant limitations in social participation.
  Measurements were conducted throughout the study, with scores compared between baseline and 8 weeks to assess changes in social participation.
Time Frame: Assessed weekly, change from baseline and Week 8 reported
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | TMC-CP01 Intervention | Standard of Care
Number analyzed (Participants) | 10 | 10
T-score | 1.95 (5) | 0.04 (4.23)

12. Secondary Outcome: Change From Baseline in Depression Using the PROMIS Short Form at 8 Weeks
Description: The investigators used the PROMIS Depression Short Form to assess depressive symptoms. This measure includes 4 items, each rated on a 5-point Likert scale (1 = never, 5 = always). The raw score (range: 4 to 20) was converted to a T-score (mean = 50, SD = 10).
  Higher T-scores indicate greater levels of depression (worse outcomes), while lower scores reflect fewer depressive symptoms. A T-score above 60 suggests clinically significant depression, while a T-score below 50 reflects better mental health relative to the general population.
  Measurements were conducted throughout the study, with scores compared between baseline and 8 weeks to assess changes in depressive symptoms.
Time Frame: Assessed weekly, change from baseline and Week 8 reported
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | TMC-CP01 Intervention | Standard of Care
Number analyzed (Participants) | 10 | 10
T-score | -1.08 (4.21) | -3.22 (6.35)

13. Secondary Outcome: Change From Baseline in Anxiety Using the PROMIS Short Form at 8 Weeks
Description: The investigators used the PROMIS Anxiety Short Form to assess anxiety symptoms. This measure includes 4 items, each rated on a 5-point Likert scale (1 = never, 5 = always). The raw score (range: 4 to 20) was converted to a T-score (mean = 50, SD = 10).
  Higher T-scores indicate greater levels of anxiety (worse outcomes), while lower scores reflect reduced anxiety symptoms. A T-score above 60 suggests clinically significant anxiety, while a T-score below 50 reflects better emotional health relative to the general population.
  Measurements were conducted throughout the study, with scores compared between baseline and 8 weeks to assess changes in anxiety symptoms.
Time Frame: Assessed weekly, change from baseline and Week 8 reported
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | TMC-CP01 Intervention | Standard of Care
Number analyzed (Participants) | 10 | 10
T-score | -4.05 (7.79) | -2.62 (5.59)

14. Secondary Outcome: Change From Baseline in Loneliness Using the PROMIS Emotional Support Short Form at 8 Weeks
Description: The investigators used the PROMIS Emotional Support Short Form to assess patient-centered outcomes related to loneliness. This measure includes 4 items, each rated on a 5-point Likert scale (1 = never, 5 = always). The raw score (range: 4 to 20) was converted to a T-score (mean = 50, SD = 10).
  Higher T-scores indicate greater loneliness (worse outcomes), while lower scores suggest better emotional support. A T-score above 60 suggests clinically significant loneliness, while a T-score below 50 reflects better perceived emotional support relative to the general population.
  Measurements were conducted throughout the study, with scores compared between baseline and 8 weeks to assess changes in loneliness.
Time Frame: Assessed weekly, change from baseline and Week 8 reported
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | TMC-CP01 Intervention | Standard of Care
Number analyzed (Participants) | 10 | 10
T-score | -2 (4.08) | -4 (5.66)

15. Secondary Outcome: Assessment of Feelings About Pain
Description: The investigators will use the PainDetect Questionnaire, a validated tool to assess patients' perceptions and feelings about pain. The questionnaire includes 15 multiple-choice questions and a drawing of localized pain, yielding a total score that ranges from 0 (minimum) to 38 (maximum). Lower scores indicate less neuropathic pain and suggest better outcomes.
Time Frame: Week 0
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TMC-CP01 Intervention | Standard of Care
Number analyzed (Participants) | 10 | 10
score on a scale | 16.9 (9.57) | 16.8 (10.73)

16. Secondary Outcome: Assessment of Feelings About Pain
Description: as for outcome 15
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TMC-CP01 Intervention | Standard of Care
Number analyzed (Participants) | 10 | 10
score on a scale | 16.89 (7.06) | 17 (5.29)

17. Secondary Outcome: Assessment of Feelings About Pain
Description: as for outcome 15
Time Frame: Week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TMC-CP01 Intervention | Standard of Care
Number analyzed (Participants) | 10 | 10
score on a scale | 14.9 (8.16) | 16.5 (8.04)

18. Secondary Outcome: Assessment of Salivary Cortisol Levels
Description: The investigators will measure subjects' salivary cortisol levels using validated laboratory techniques. Cortisol levels are reported in micrograms per deciliter (mcg/dL) and have no predefined minimum or maximum values. Lower cortisol levels indicate better outcomes.
Time Frame: Week 0
Measure: Mean (Standard Deviation); unit: mcg/dL
Arm/Group | TMC-CP01 Intervention | Standard of Care
Number analyzed (Participants) | 10 | 10
mcg/dL | 3.68 (2.32) | 5.07 (5.06)

19. Secondary Outcome: Assessment of Salivary Cortisol Levels
Description: as for outcome 18
Time Frame: Week 4
Population: Data were not collected at Week 4 because salivary cortisol levels were only measured at baseline (Week 0) and the study endpoint (Week 8). No data exist for this time point.
Arm/Group | TMC-CP01 Intervention | Standard of Care
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Assessment of Salivary Cortisol Levels
Description: as for outcome 18
Time Frame: Week 8
Measure: Mean (Standard Deviation); unit: mcg/dL
Arm/Group | TMC-CP01 Intervention | Standard of Care
Number analyzed (Participants) | 10 | 10
mcg/dL | 6.72 (5.73) | 8.38 (9.15)

21. Secondary Outcome: Assessment of Opioid Use Via Urinalysis
Description: The amount of opiates found in the urine of each subject will be recorded throughout the study. The lower the detected morphine milligram equivalent [MME], the better the outcomes. Outcomes will be measured over the span of the study and compared between the two groups.
Time Frame: Week 0
Population: Urine drug screen data were not collected due to two key barriers: (1) the clinical personnel required to administer the tests were not consistently available during study visits, and (2) the cost of performing quantitative urine drug screens for each participant was beyond the scope of the study's budget. As a result, no data are available for this outcome.
Arm/Group | TMC-CP01 Intervention | Standard of Care
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: Assessment of Opioid Use Via Urinalysis
Description: as for outcome 21
Time Frame: Week 4
Population: as for outcome 21
Arm/Group | TMC-CP01 Intervention | Standard of Care
Number analyzed (Participants) | 0 | 0

23. Secondary Outcome: Assessment of Opioid Use Via Urinalysis
Description: as for outcome 21
Time Frame: Week 8
Population: as for outcome 21
Arm/Group | TMC-CP01 Intervention | Standard of Care
Number analyzed (Participants) | 0 | 0

24. Secondary Outcome: Assessment of Withdrawal Symptoms Using Opiate Withdrawal Scale
Description: The Subjective Opiate Withdrawal Scale (SOWS) will assess subjects' withdrawal symptoms using 16 multiple-choice questions, each scored from 0 (not at all) to 4 (extremely). The total score ranges from a minimum of 0 to a maximum of 64. Lower scores indicate better outcomes and fewer withdrawal symptoms.
Time Frame: Week 0
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TMC-CP01 Intervention | Standard of Care
Number analyzed (Participants) | 10 | 10
score on a scale | 8 (5.37) | 3.7 (2.83)

25. Secondary Outcome: Assessment of Withdrawal Symptoms Using Opiate Withdrawal Scale
Description: as for outcome 24
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TMC-CP01 Intervention | Standard of Care
Number analyzed (Participants) | 10 | 10
score on a scale | 7.67 (4.82) | 14 (18.52)

26. Secondary Outcome: Assessment of Withdrawal Symptoms Using Opiate Withdrawal Scale
Description: as for outcome 24
Time Frame: Week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TMC-CP01 Intervention | Standard of Care
Number analyzed (Participants) | 10 | 10
score on a scale | 7.6 (6.35) | 5.67 (6.92)

27. Secondary Outcome: Assessment of Beliefs About Pain Using Pain Catastrophizing Scale
Description: The Pain Catastrophizing Scale (PCS) will assess subjects' beliefs about pain using 13 multiple-choice questions, each scored from 1 (not at all) to 5 (all the time). The total score ranges from a minimum of 13 to a maximum of 65. Lower scores indicate better outcomes and less catastrophizing about pain.
Time Frame: Week 0
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TMC-CP01 Intervention | Standard of Care
Number analyzed (Participants) | 10 | 10
score on a scale | 31.33 (9.12) | 25.8 (10.9)

28. Secondary Outcome: Assessment of Beliefs About Pain Using Pain Catastrophizing Scale
Description: as for outcome 27
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TMC-CP01 Intervention | Standard of Care
Number analyzed (Participants) | 10 | 10
score on a scale | 34.4 (10.01) | 25.29 (7.54)

29. Secondary Outcome: Assessment of Beliefs About Pain Using Pain Catastrophizing Scale
Description: as for outcome 27
Time Frame: Week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TMC-CP01 Intervention | Standard of Care
Number analyzed (Participants) | 10 | 10
score on a scale | 27.1 (9.48) | 23.71 (7.83)

30. Secondary Outcome: Assessment of Treatment Expectancy Using the Treatment Expectancy Short Form at Week 0
Description: The Treatment Expectancy Short Form assesses subjects' expectations and confidence in their treatment using 6 items, each scored on a 5-point Likert scale (1 = not at all, 5 = very much). The raw score (range: 6 to 30) is converted to a T-score (mean = 50, SD = 10) for standardized interpretation.
  Higher T-scores indicate greater treatment expectancy, suggesting more positive beliefs about treatment efficacy. Lower T-scores reflect greater skepticism or uncertainty. A T-score above 60 may indicate high confidence in treatment, while a T-score below 40 suggests low expectancy.
Time Frame: Week 0
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | TMC-CP01 Intervention | Standard of Care
Number analyzed (Participants) | 10 | 10
t-score | 50.19 (6.03) | 51.33 (5.7)

31. Secondary Outcome: Assessment of Treatment Expectancy Using the Treatment Expectancy Short Form at Week 4
Description: as for outcome 30
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | TMC-CP01 Intervention | Standard of Care
Number analyzed (Participants) | 10 | 10
t-score | 46.04 (6.95) | 51.43 (5.45)

32. Secondary Outcome: Assessment of Treatment Expectancy Using the Treatment Expectancy Short Form at Week 8
Description: The Treatment Expectancy Short Form evaluates subjects' expectations and confidence in their treatment using 6 items, each rated on a 5-point Likert scale (1 = not at all, 5 = very much). The raw score (range: 6 to 30) is converted to a T-score (mean = 50, SD = 10) for standardized interpretation.
  Higher T-scores indicate greater treatment expectancy, suggesting more positive beliefs about treatment efficacy. Lower T-scores reflect greater skepticism or uncertainty. A T-score above 60 may indicate high confidence in treatment, while a T-score below 40 suggests low expectancy.
Time Frame: Week 8
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | TMC-CP01 Intervention | Standard of Care
Number analyzed (Participants) | 10 | 10
T-score | 50.48 (8.65) | 43.98 (10.21)

33. Secondary Outcome: Assessment of Positive Outlook Using the Positive Outlook Short Form at Week 0
Description: The Positive Outlook Short Form measures subjects' perceptions and feelings about the future using 6 items, each rated on a 5-point Likert scale (1 = not at all, 5 = very much). The raw score (range: 6 to 30) is converted to a T-score (mean = 50, SD = 10) for standardized interpretation.
  Higher T-scores indicate greater optimism and a more positive outlook, suggesting better psychological well-being. Lower T-scores reflect greater pessimism or concerns about the future. A T-score above 60 may indicate high optimism, while a T-score below 40 suggests low optimism or increased negative expectations.
Time Frame: Week 0
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | TMC-CP01 Intervention | Standard of Care
Number analyzed (Participants) | 10 | 10
T-score | 46.06 (9.53) | 50.22 (11.77)

34. Secondary Outcome: Assessment of Positive Outlook Using the Positive Outlook Short Form at Week 4
Description: as for outcome 33
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | TMC-CP01 Intervention | Standard of Care
Number analyzed (Participants) | 10 | 10
T-score | 46.77 (6.47) | 53.43 (17.6)

35. Secondary Outcome: Assessment of Positive Outlook Using the Positive Outlook Short Form at Week 8
Description: The Positive Outlook Short Form evaluates subjects' perceptions and expectations about the future using 6 items, each rated on a 5-point Likert scale (1 = not at all, 5 = very much). The raw score (range: 6 to 30) is converted to a T-score (mean = 50, SD = 10) for standardized interpretation.
  Higher T-scores indicate greater optimism and a more positive outlook, suggesting better psychological well-being. Lower T-scores reflect greater pessimism or concerns about the future. A T-score above 60 may indicate high optimism, while a T-score below 40 suggests low optimism or increased negative expectations.
Time Frame: Week 8
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | TMC-CP01 Intervention | Standard of Care
Number analyzed (Participants) | 10 | 10
T-score | 46.86 (8.89) | 50.48 (12.21)

36. Secondary Outcome: Assessment of Recent Behaviors Using the Current Opioid Misuse Measure (COMM)
Description: The Current Opioid Misuse Measure (COMM) questionnaire assesses recent behaviors using 17 multiple-choice questions, with scores ranging from a minimum of 0 to a maximum of 68. Lower scores suggest better outcomes and less likelihood of opioid misuse.
Time Frame: Week 0
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TMC-CP01 Intervention | Standard of Care
Number analyzed (Participants) | 10 | 10
score on a scale | 11 (6.07) | 9 (5.93)

37. Secondary Outcome: Assessment of Recent Behaviors Using the Current Opioid Misuse Measure (COMM)
Description: as for outcome 36
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TMC-CP01 Intervention | Standard of Care
Number analyzed (Participants) | 10 | 10
score on a scale | 7.89 (5.78) | 6 (2)

38. Secondary Outcome: Assessment of Recent Behaviors Using the Current Opioid Misuse Measure (COMM)
Description: as for outcome 36
Time Frame: Week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TMC-CP01 Intervention | Standard of Care
Number analyzed (Participants) | 10 | 10
score on a scale | 10.10 (7.36) | 3.17 (2.93)

39. Secondary Outcome: Assessment of Task Absorption Using the Tellegen Absorption Scale (TAS) at Week 0
Description: The Tellegen Absorption Scale (TAS) assesses an individual's ability to become deeply engaged in a task or an aspect of their environment. The scale consists of 34 true-or-false items, where each "true" response is scored as 1, and each "false" response is scored as 0.
  The total score ranges from 0 to 34, with higher scores indicating a greater capacity for absorption and immersive engagement. This measure evaluates attentional focus and deep engagement in activities, which may be relevant for assessing response to virtual reality interventions.
Time Frame: Week 0
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | TMC-CP01 Intervention | Standard of Care
Number analyzed (Participants) | 10 | 10
Units on a scale | 10.2 (7.41) | 14.3 (8.53)

40. Secondary Outcome: Assessment of Task Absorption Using the Tellegen Absorption Scale (TAS) at Week 4
Description: as for outcome 39
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | TMC-CP01 Intervention | Standard of Care
Number analyzed (Participants) | 10 | 10
Units on a scale | 9.22 (8.15) | 17.67 (8.02)

41. Secondary Outcome: Assessment of Task Absorption Using the Tellegen Absorption Scale (TAS) at Week 8
Description: as for outcome 39
Time Frame: Week 8
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | TMC-CP01 Intervention | Standard of Care
Number analyzed (Participants) | 10 | 10
Units on a scale | 8.4 (7.15) | 16 (7.92)

42. Secondary Outcome: Change in Pain Level Before vs After Intervention Via Flowly App
Description: Subjects rated their current pain level using the 0-10 Visual Analog Scale (VAS) within the Flowly app, where 0 represents no pain and 10 represents the worst imaginable pain. Pain scores were recorded immediately before and after each VR session, which took place daily throughout the study.
  For analysis, pain scores were assessed at baseline and at Week 8. The Week 8 value represents the average of daily post-session scores recorded during the final week of the study. The change in pain levels was calculated by comparing the baseline value to the Week 8 average.
  Higher scores indicate greater pain intensity, while lower scores suggest better outcomes (i.e., pain reduction).
Time Frame: Baseline and Week 8 (Week 8 value is the average of daily scores from that week)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | TMC-CP01 Intervention | Standard of Care
Number analyzed (Participants) | 10 | 10
Units on a scale | 0.2 (1.32) | 0.14 (1.07)

43. Secondary Outcome: Change in Anxiety Level From Baseline to 8 Weeks Via Flowly App
Description: Subjects rated their current anxiety level using the 0-10 Visual Analog Scale (VAS) within the Flowly app, where 0 represents no anxiety and 10 represents the worst imaginable anxiety. Anxiety scores were recorded immediately before and after each VR session, which took place daily throughout the study.
  For analysis, anxiety scores were assessed at baseline and at Week 8. The Week 8 value represents the average of daily post-session scores recorded during the final week of the study. The change in anxiety levels was calculated by comparing the baseline value to the Week 8 average.
  Higher scores indicate greater anxiety levels, while lower scores suggest better outcomes (i.e., anxiety reduction).
Time Frame: Baseline and Week 8 (Week 8 value is the average of daily scores from that week)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | TMC-CP01 Intervention | Standard of Care
Number analyzed (Participants) | 10 | 10
Units on a scale | -4.05 (7.79) | -2.62 (5.59)

44. Secondary Outcome: Change in Depression Level From Baseline to 8 Weeks Via Flowly App
Description: Subjects rated their current depression level using the 0-10 Visual Analog Scale (VAS) within the Flowly app, where 0 represents no depression and 10 represents the worst imaginable depression. Depression scores were recorded immediately before and after each VR session, which took place daily throughout the study.
  For analysis, depression scores were assessed at baseline and at Week 8. The Week 8 value represents the average of daily post-session scores recorded during the final week of the study. The change in depression levels was calculated by comparing the baseline value to the Week 8 average.
  Higher scores indicate greater depression levels, while lower scores suggest better outcomes (i.e., depression reduction).
Time Frame: Baseline and Week 8 (Week 8 value is the average of daily scores from that week)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | TMC-CP01 Intervention | Standard of Care
Number analyzed (Participants) | 10 | 10
Units on a scale | -1.08 (4.21) | -3.22 (6.35)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from baseline to study completion (8 weeks).
Arm/Group | TMC-CP01 Intervention | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

LIMITATIONS AND CAVEATS:
The primary limitation of this study is the small sample size (n=20), which may impact statistical power and generalizability. While analyses were conducted, the limited number of participants affects the ability to detect statistically significant differences or draw broader conclusions. Larger trials are necessary to further evaluate the intervention's effects and determine its reproducibility in a larger population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-12-20): https://cdn.clinicaltrials.gov/large-docs/04/NCT04236804/Prot_SAP_001.pdf
  • Informed Consent Form (2021-04-20): https://cdn.clinicaltrials.gov/large-docs/04/NCT04236804/ICF_000.pdf